CLINICAL TRIAL: NCT06045637
Title: The Effect of Cognitive Behavioral Approach-based Psychoeducation on the Cognitive Emotion Regulation Strategies and Negative Emotional Symptom Levels of Emerging Adults Who Experienced an Earthquake
Brief Title: The Effect of Psychoeducation on Cognitive Emotion Regulation and Negative Emotional Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Ahmet Çapar, Principal Investigator, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OKU-SBF-AC-01
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Earthquake
Keywords: emerging adulthood; cognitive emotion regulation; negative emotional symptoms; psychoeducation; cognitive behavioral approach

STUDY DESIGN:
Intervention Model Description: This research was planned as a randomized controlled experimental study. In this research, pre-test, post-test and follow-up test will be performed and there will be 1 experimental and 1 control group created by randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group included in a psychoeducational program based on cognitive behavioral approach (experiment) (Experimental): Emerging adults between the ages of 18-29 who experienced the Kahramanmaraş 2023 earthquake in Turkey constitute the experimental group.
  The cognitive behavioral approach-based psychoeducation program will be implemented in 9 sessions, two days a week and 90 minutes a day.In the psychoeducation program, based on the cognitive behavioral approach, trauma and trauma symptoms, emotion-thought-behavior analysis, cognitive errors, automatic thoughts, alternative thought generation, mentality and distorted thoughts that reveal feelings of depression, anxiety, stress, anger, guilt, inadequacy, helplessness, The cognitive aspect of hopelessness and methods of coping with negative emotions will be discussed.The training program includes verbal expression, visual material (projection), question and answer, homework, sample stories, entertaining activities, warm-up games, etc. It will be continued and feedback will be shared.
  Interventions: Behavioral: Group included in a psychoeducational program based on the cognitive behavioral approach (experiment)
- Group not included in the psychoeducation program based on cognitive behavioral approach (Control) (No Intervention): No intervention will be made to this group.

INTERVENTIONS:
Behavioral: Group included in a psychoeducational program based on the cognitive behavioral approach (experiment) — The 9-session cognitive behavioral approach-based psychoeducation program will last 5 weeks. Sessions; It will be carried out in the form of acquaintance, recognition of trauma and its effects, emotion and thought behavior analysis, cognitive errors, automatic thoughts and alternative thought generation, cognitive emotion regulation strategies, coping with negative emotions, instilling hope and termination session.
  Arms: Group included in a psychoeducational program based on cognitive behavioral approach (experiment)

SUMMARY:
This research was planned to determine the effect of cognitive behavioral approach-based psychoeducation on the cognitive emotion regulation strategies and negative emotional symptom levels of emerging adults who experienced an earthquake. In this research, pre-test, post-test and follow-up test will be performed and there will be 1 experimental and 1 control group created by randomization.After the pre-test applied to the experimental and control groups, a 9-session cognitive behavioral approach-based psychoeducation program will be applied to the experimental group.Following this application, post-test and one-month follow-up tests will be administered to both groups and the effectiveness of the psychoeducation program will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being in the 18-29 age group,
* Being at least a primary school graduate,
* Being exposed to/having experienced the Kahramanmaraş earthquake and living in the center of Osmaniye.

Exclusion Criteria:

* Having a hearing or speech disability that makes it difficult to answer surveys,
* Participating in a similar psychoeducation program,
* Presence of any psychiatric disorder and receiving treatment

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
cognitive emotion regulation scale | Two months
  The scale consists of 36 items, with 9 subscales and 4 items in each subscale. Each subscale receives a value between 4-20 points and the scale is a 5-point Likert type scale (1: Never, 2: Sometimes, 47 3: Regularly, 4: Frequently, 5: Always).Evaluation is made with the scores obtained from the subscales. A higher score from a subscale indicates greater use of the cognitive emotion regulation strategy determined by that subscale.
Depression, Anxiety, Stress Scale | Two months
  The scale consists of 21 items, with 3 sub-dimensions (depression, anxiety and stress) and 7 items in each sub-dimension.
  The scale is designed as a self-evaluation scale with a 4-point Likert structure scored between 0-4. (0- Never, 1- Sometimes and occasionally, 2- Quite often, 3- Always). The scoring range of the scale for depression is: 0-4 normal, 5-6 mild, 7-10 moderate, 11-13 severe, 14 and above very severe; for anxiety: 0-3 normal, 4-5 mild, 6-7 moderate, 8-9 severe, and 10 and above very severe; For stress: 0-7 is normal, 8-9 is mild, 10-12 is moderate, 13-16 is severe, 17 and above is very severe.

CONTACTS AND LOCATIONS:
Overall Officials: AHMET ÇAPAR, lecturer, Principal Investigator — Osmaniye Korkut Ata University
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No